CLINICAL TRIAL: NCT04330794
Title: the NMFACT Anew Caries Index
Brief Title: the NMFACT Caries Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 23456
Record Dates: First submitted 2018-07-16; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — DMF Index

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMFACT (Experimental): record the caries index using the NMFACT chart
  Interventions: Other: NMFACT
- DMF index (Active Comparator): record the caries index using the DMF chart
  Interventions: Other: DMF index

INTERVENTIONS:
Other: NMFACT — caries index
  Other Names: NMFACT chart
  Arms: NMFACT
Other: DMF index — caries index chart to collect data about decayed missed filled teeth
  Other Names: DMF chart
  Arms: DMF index

SUMMARY:
the NMFACT is a new caries index to overcome the drawbacks of DMF cries index the ''N'' is for non carious lesion, the ''M''for missed teeth,the ''F''for filled teeth,the''C''for carious teeth,the ''A''for alignment and the ''T''for dental trauma.

each problem will be scored from 0(normal).

DETAILED DESCRIPTION:
the new caries index will be used to record the dental problem . the validation will be recorded against the gold standard DMF index

ELIGIBILITY:
Inclusion Criteria:

* any patient suffering form dental problem

Exclusion Criteria:

* edentulous patient children adolescents

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
the accuracy of NMFACT index in describe the oral health condition | 3months
  finding from the group will be compared to clinical examination by different accessors .the accurate detailed description of the oral health condition will assessed statistically

IPD SHARING:
Plan to Share IPD: No